CLINICAL TRIAL: NCT04401293
Title: Systemic Anticoagulation With Full Dose Low Molecular Weight Heparin (LMWH) Vs. Prophylactic or Intermediate Dose LMWH in High Risk COVID-19 Patients (HEP-COVID Trial)
Brief Title: Full Dose Heparin Vs. Prophylactic Or Intermediate Dose Heparin in High Risk COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Alex Spyropoulos, System Director - Anticoagulation and Clinical Thrombosis Services Northwell Health at Lenox Hill Hospital, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0340
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Sars-CoV2; COVID
Keywords: COVID-19; Anticoagulation; Heparin; Coronavirus; Thrombosis
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Thrombosis | interventions — Enoxaparin; Heparin; Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Due to the pragmatic nature of this study "open-label multi-center randomized active control trial" with pseudo-blinding mechanisms at the time of randomization the study subject and corresponding Site PIs will be blinded (unaware of specific treatment arm the patient is assigned to i.e. Arm 0 or Arm 1). The study pharmacists as well as data extractors and designated randomization personnel (i.e. research coordinators and/or research nurses performing the randomization process) will be un-blinded (aware of specific treatment arm the patient is assigned to i.e. Arm 0 or Arm 1). At the time of subject randomization study subjects will be stratified to either ICU level of care vs. Non-ICU level of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full Dose LMWH anticoagulation therapy (Experimental): Subjects in this study arm will be treated with therapeutic doses of subcutaneous low-molecular-weight heparin (enoxaparin). Enoxaparin 1mg/kg SQ BID for CrCl ≥ 30ml/min (or Enoxaparin 0.5mg/kg SQ BID for CrCl ≥ 15ml/min and < 30ml/min) during the course of their hospitalization.
  Interventions: Drug: Enoxaparin
- Prophylactic/Intermediate Dose LMWH or UFH therapy (Active Comparator): Subjects in this study arm will be treated with Local institutional standard-of-care for prophylactic-dose or intermediate-dose UFH or LMWH. Regimens allowed are UFH up to 22,500 IU daily in BID or TID doses (i.e. UFH 5000 IU SQ BID/TID or 7500 IU BID/TID), enoxaparin 30mg and 40mg SQ QD or BID (the use of weight-based enoxaparin i.e. 0.5mg/kg SQ BID for this arm is acceptable but strongly discouraged), dalteparin 2500IU or 5000IU QD.
  Interventions: Drug: Prophylactic/Intermediate Dose Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Full Dose LMWH anticoagulation therapy
  Arms: Full Dose LMWH anticoagulation therapy
Drug: Prophylactic/Intermediate Dose Enoxaparin — Prophylactic/Intermediate Dose LMWH or UFH therapy
  Other Names: Unfractionated heparin; dalteparin
  Arms: Prophylactic/Intermediate Dose LMWH or UFH therapy

SUMMARY:
The aim of this study is to test the hypothesis that prophylaxis of severe COVID-19 patients with treatment dose LMWH leads to better thromboembolic-free outcomes and associated complications during hospitalization than prophylaxis with institutional standard of care with prophylactic to intermediate-doses of UFH or LMWH

DETAILED DESCRIPTION:
There are clinical data to support the observation that hospitalized acutely ill medical patients with severe viral pneumonitis/Acute Respiratory Distress Syndrome (ARDS), such as those with influenza H1N1 infection, have an over 23-fold increased risk for venous thromboembolism (VTE) - especially pulmonary embolism (PE) - with an overall 44% incidence of VTE in ARDS associated with H1N1 pneumonia. Multicenter studies from China report that key markers of inflammation and/or coagulopathy are associated with morbidity and increased mortality in COVID-19 patients. Elevated D-dimer levels (that are sometime greater than 4 or 6 times the upper limit of normal [ULN]) are strongly associated with mortality in patients with severe COVID-19 illness. Recent data also shows that mortality among COVID-19 patients is markedly higher in patients with elevated Troponin-T (TnT) levels than in patients with normal TnT levels. Recently a cohort of 81 patients retrospectively evaluated diagnosed with severe COVID-19 pneumonia and reported a lower extremity VTE incidence of 25% (20/81) and a mortality of 40% (8/20) in the presence of VTE. Reported a case of bilateral pulmonary embolism in a 75 year old woman diagnosed with severe COVID-19, in the absence of predisposing risk factors and a negative lower extremity US. Lastly the investigated use of Tissue Plasminogen Activator (tPA) in the treatment of COVID-19 associated ARDS and reported promising, but transient, results in terms of pulmonary function improvement. It appears that either the SARS-CoV2 infection itself induces a hypercoagulable state, possibly by hypofibrinolytic mechanisms, or the cytokine storm in COVID-19 patients with severe disease induces a prothrombotic state, which leads to clinical deterioration, hypoxia and hemodynamic instability secondary to thromboembolic phenomena and potentially cardiac ischemia. Preliminary data from Northwell Health System, which has one of the largest populations of hospitalized COVID-19 patients in the US, reveals a positivity rate for deep vein thrombosis (DVT) of 40% of those COVID-19 patients screened by Doppler compression ultrasonography of the lower extremities.

Heparin has been shown to have anti-inflammatory and immunomodulatory properties in addition to its anticoagulation effect, which could play a beneficial role in sepsis. In addition, there is in vitro evidence that the large negatively charged sulfated glycosaminoglycans of unfractionated heparin may act as an alternate ligand for the SARS-CoV2 receptor irrespective of ACE2. Whether this in vitro evidence supports the role of a protective or deleterious mechanism in COVID-19 infection is not known. However, an early report with empiric use of treatment dose unfractionated heparin (UFH) in ARDS from a different viral family, influenza H1N1, revealed that H1N1 ARDS patients under systemic anticoagulation had 33-fold fewer VTE events than those treated given prophylactic doses of UFH/low-molecular weight heparin (LMWH) thromboprophylaxis. Very recent evidence suggests that therapy with prophylactic to intermediate doses of the LMWH enoxaparin (30mg to 60mg QD) in severe hospitalized COVID-19 patents with a SIC score ≥ 4 or D-dimer (Dd) > 6 X ULN improves outcomes and prognosis. All-cause mortality at 28 days was reduced from 64.2% to 40.0% in those patients with a SIC score ≥ 4 (p=0.029), and from 52.4% to 32.8% in those patients with an elevated Dd > 6 x ULN (P=0.017). Notably, Klok and colleagues investigated 184 ICU patients infected with COVID-19 and reported a 13% mortality rate, a relatively high incidence of CTPA- or ultrasonography-confirmed VTE rate (27%), and arterial thrombotic events (3.7%) despite the use of standard dose thromboprophylaxis. Postulated mechanisms for the improved prognosis with the use of treatment doses of LMWH in the sick COVID-19 population include the decrease in the risk of microthrombi, especially in the pulmonary vasculature, which can lead to hypoxemia, pulmonary vasoconstriction and right ventricular dysfunction as well as the decrease in the risk of progression to disseminated intravascular coagulopathy as a contributor to the high mortality seen in these patients.

The optimal dose of heparin (either LMWH or UFH) in hospitalized COVID-19 patients is unknown, as patients on conventional prophylactic dose heparin (UFH or LMWH) as supported by international guidance statements on hospitalized COVID-19 patients appear to remain at risk for thromboembolic events. There is data to support improved efficacy with treatment doses of twice daily enoxaparin versus once-daily weight-adjusted enoxaparin for the management of VTE, especially with large thrombus burden. There is also long-standing data to support that treatment-dose heparin can reduce major cardiovascular events. Our current standard of care in our 24 hospital Northwell Health System, which has a very large hospitalized COVID-19 patient population, is to use Lovenox 40mg SQ QD for patients with a BMI < 30 and Creatinine Clearance (CrCl) > 15ml/min, Lovenox 40mg SQ BID for patients with a BMI > 30 and CrCl > 15ml/min, and UFH 5000U SQ BID or TID in patients with a CrCl < 15ml/min and BMI < 30 and UFH 7500U SQ BID or TID with a CrCl < 15ml/min and BMI > 30. Large healthcare institutions in the US and elsewhere have protocols for in-patient thromboprophylaxis ranging from prophylactic-to-intermediate dose UFH or LMWH for the management of patients with COVID-19 associated coagulopathy. The aim of this study is to test the hypothesis that prophylaxis of severe COVID-19 patients with treatment dose LMWH leads to better thromboembolic-free outcomes and associated complications during hospitalization than prophylaxis with institutional standard of care with prophylactic to intermediate-doses of UFH or LMWH.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
2. Understands and agrees to comply with planned study procedures.
3. Male or non-pregnant female adult ≥18 years of age at time of enrollment.
4. Subject consents to randomization within 72 hours of hospital admission or transfer from another facility within 72 hours of index presentation.
5. Subjects with a positive COVID-19 diagnosis by nasal swab or serologic testing.
6. Hospitalized with a requirement for supplemental oxygen.
7. Have:

   * Either a D- Dimer > 4.0 X ULN, OR
   * Sepsis-induced coagulopathy (SIC) score of ≥4

Exclusion Criteria:

1. Indications for therapeutic anticoagulation
2. Absolute contraindication to anticoagulation including:

   1. active bleeding,
   2. recent (within 1 month) history of bleed,
   3. dual (but not single) antiplatelet therapy,
   4. active gastrointestinal and intracranial cancer,
   5. a history of bronchiectasis or pulmonary cavitation,
   6. Hepatic failure with a baseline INR > 1.5,
   7. CrCl < 15ml/min,
   8. a platelet count < 25,000,
   9. a history of heparin-induced thrombocytopenia (HIT) within the past 100 days or in the presence of circulating antibodies,
   10. contraindications to enoxaparin including a hypersensitivity to enoxaparin sodium, hypersensitivity to heparin or pork products, hypersensitivity to benzyl alcohol,
   11. pregnant female,
   12. inability to give or designate to give informed consent,
   13. participation in another blinded trial of investigational drug therapy for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2020-04-26 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex C Spyropoulos, MD, Principal Investigator — Northwell Health
Locations (6):
- United States (6):
  - Beth Israel Newark, Newark, New Jersey
  - Southside Hospital, Bay Shore, New York
  - Huntington Hospital, Huntington, New York
  - Lenox Hill Hospital, New York, New York
  - Long Island Jewish Medical Center, Queens, New York
  - Staten Island University Hospital, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Spyropoulos AC, Goldin M, Giannis D, Diab W, Wang J, Khanijo S, Mignatti A, Gianos E, Cohen M, Sharifova G, Lund JM, Tafur A, Lewis PA, Cohoon KP, Rahman H, Sison CP, Lesser ML, Ochani K, Agrawal N, Hsia J, Anderson VE, Bonaca M, Halperin JL, Weitz JI; HEP-COVID Investigators. Efficacy and Safety of Therapeutic-Dose Heparin vs Standard Prophylactic or Intermediate-Dose Heparins for Thromboprophylaxis in High-risk Hospitalized Patients With COVID-19: The HEP-COVID Randomized Clinical Trial. JAMA Intern Med. 2021 Dec 1;181(12):1612-1620. doi: 10.1001/jamainternmed.2021.6203. PMID 34617959
- [Derived] Short SAP, Gupta S, Brenner SK, Hayek SS, Srivastava A, Shaefi S, Singh H, Wu B, Bagchi A, Al-Samkari H, Dy R, Wilkinson K, Zakai NA, Leaf DE; STOP-COVID Investigators. d-dimer and Death in Critically Ill Patients With Coronavirus Disease 2019. Crit Care Med. 2021 May 1;49(5):e500-e511. doi: 10.1097/CCM.0000000000004917. PMID 33591017
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773
- See also: Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the Coronavirus Disease 2019 (COVID-19) Pandemic — https://doi.org/10.1016/j.jacc.2020.03.031
- See also: Empirical systemic anticoagulation is associated with decreased venous thromboembolism in critically ill influenza A H1N1 acute respiratory distress syndrome patients — https://doi.org/10.1016/j.jvsv.2018.08.010
- See also: Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia — https://doi.org/10.1111/jth.14768
- See also: Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy — https://doi.org/10.1111/jth.14817
- See also: Prevalence of venous thromboembolism in patients with severe novel coronavirus pneumonia — https://doi.org/10.1111/jth.14830
- See also: Tissue Plasminogen Activator (tPA) Treatment for COVID-19 Associated Acute Respiratory Distress Syndrome (ARDS): A Case Series — https://doi.org/10.1111/jth.14828
- See also: Pharmacology of Heparin and Related Drugs — https://doi.org/10.1124/pr.115.011247
- See also: Incidence of thrombotic complications in critically ill ICU patients with COVID-19 — https://doi.org/10.1016/j.thromres.2020.04.013
- See also: Bivalirudin or Heparin in Patients Undergoing Invasive Management of Acute Coronary Syndromes — https://doi.org/10.1016/j.jacc.2018.01.033
- See also: Emergence of Institutional Antithrombotic Protocols for Coronavirus 2019 — https://doi.org/10.1002/rth2.12358

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Started | 130 | 127
Completed | 129 | 124
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy | Total
Number analyzed (Participants) | 129 | 124 | 253
Age, Customized [Mean (Standard Deviation); unit: years]
  Age in Years | 65.8 (13.9) | 67.7 (14.1) | 66.7 (14.00)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 68 | 68 | 136
  Female | 61 | 56 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 14 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 37 | 70
  White | 56 | 46 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome of Arterial Thromboembolic Events, Venous Thromboembolic Events and All-cause Mortality at Day 30 ± 2 Days.
Description: Risk of arterial thromboembolic events (including myocardial infarction, stroke, systemic embolism), venous thromboembolism (including symptomatic deep vein thrombosis (DVT) of the upper or lower extremity, asymptomatic proximal DVT of the lower extremity, non-fatal pulmonary embolism (PE)), and all-cause mortality at Day 30 ± 2 days.
Time Frame: Day 30 ± 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Number analyzed (Participants) | 129 | 124
Participants | 25 | 31

2. Secondary Outcome: Major Bleeding
Description: Risk of major bleeding defined using the International Society of Thrombosis and Haemostasis (ISTH) criteria
Time Frame: Day 30 ± 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Number analyzed (Participants) | 129 | 124
Participants | 6 | 2

3. Secondary Outcome: Composite Outcome of Arterial Thromboembolic Events, Venous Thromboembolic Events and All-cause Mortality at Hospital Day 10 + 4
Description: The composite of arterial thromboembolic events (including myocardial infarction, stroke, systemic embolism), venous thromboembolism (including symptomatic deep vein thrombosis (DVT) of the upper or lower extremity, asymptomatic proximal DVT of the lower extremity, non-fatal pulmonary embolism (PE)), and all-cause mortality at Hospital Day 10 + 4
Time Frame: Day 10 + 4
Measure: Count of Participants; unit: Participants
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Number analyzed (Participants) | 129 | 124
Participants | 2 | 3

4. Secondary Outcome: Sepsis-induced Coagulopathy (SIC) Score
Description: Sepsis-induced coagulopathy (SIC) score predicts likelihood of sepsis-induced coagulopathy based on ISTH guidelines.
  The score uses the following domains:
  * Platelets, K/uL (thousands per microliter)
  * INR (International Normalized Ratio)
  * D-Dimer Level
  * Fibrinogen
  Platelet count > 100 cells x 10^9/L is 0 points, platelet count 50 to 100 cells x 10^9/L is 1 point and Platelet count < 50 cells x 10^9/L is 2 points. INR < 1.3 is 0 points, INR 1.3 to 1.7 is 1 point and INR > 1.7 is 2 points. D-Dimer level < 400 ng/mL is 0 points, D-Dimer level 400-4000 ng/mL is 2 points and D-Dimer level > 4000 ng/mL is 3 points. Fibrinogen level > 100 mg/dL is 0 points and fibrinogen level < 100 mg/dL is 1 point.
  Calculated (SIC) scores yields a possible 0 to 6 points, where ≥4 predicts higher mortality rates within 30 days and greater risk of pulmonary embolism.
Time Frame: Day 30 ± 2 days.
Population: COVID-19 patients have been noted to have significantly elevated markers of hypercoagulability including d-dimer (Dd), fibrinogen levels, FVIII levels, short activated partial thromboplastin time (aPTT) and Sepsis-Induced Coagulopathy (SIC) scores with an increase in venous thromboembolic disease as well as cardiac injury.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Number analyzed (Participants) | 129 | 124
units on a scale | 2.35 (0.73) | 2.31 (0.85)

5. Secondary Outcome: Progression to Acute Respiratory Distress Syndrome (ARDS)
Description: Progression to Acute Respiratory Distress Syndrome (ARDS) based on monitoring of patient conditions.
Time Frame: Day 30 ± 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Number analyzed (Participants) | 127 | 121
Participants | 11 | 6

6. Secondary Outcome: Need for Intubation
Description: Need for Intubation will be based on monitoring of patient conditions.
Time Frame: Day 30 ± 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Number analyzed (Participants) | 122 | 121
Participants | 17 | 21

7. Secondary Outcome: Re-hospitalization
Description: Need for Re-hospitalization will be based on monitoring of patient conditions.
Time Frame: Day 30 ± 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
Number analyzed (Participants) | 129 | 124
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: From screening/randomization, adverse event data was monitored and collected for each participant for 30 days (± 2 days), which was their duration in the study.
Arm/Group | Full Dose LMWH Anticoagulation Therapy | Prophylactic/Intermediate Dose LMWH or UFH Therapy
All-Cause Mortality (participants affected / at risk) | 25/129 | 31/124
Serious Adverse Events (participants affected / at risk) | 2/129 | 0/124
Other Adverse Events (participants affected / at risk) | 0/129 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Dose LMWH Anticoagulation Therapy (N=129) | Prophylactic/Intermediate Dose LMWH or UFH Therapy (N=124)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Patient was found to have low platelets during this admission. Low platelets were probably due to the blood thinner she was taking (lovenox). Excessive bruising and ecchymosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT04401293/Prot_SAP_003.pdf
  • Informed Consent Form (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT04401293/ICF_004.pdf